CLINICAL TRIAL: NCT03874013
Title: A Phase 3, Open-Label, Randomized, Multicenter, 12-month, Efficacy and Safety Study of Weekly MOD-4023 Compared to Daily Genotropin® Therapy in Japanese Pre-pubertal Children With Growth Hormone Deficiency
Brief Title: Safety and Efficacy Study of MOD-4023 to Treat Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CP-4-009
Record Dates: First submitted 2018-10-01; First posted 2019-03-14 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — MOD-4023; somatrogon; Human Growth Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MOD-4023 Treatment Arm (Experimental): MOD-4023 (investigational treatment): weekly MOD-4023 SC injections for 12 months; initially over the first 6 weeks, MOD-4023 will be administered in 3 stepwise escalating doses (0.25 mg/kg/week, 0.48 mg/kg/week and 0.66 mg/kg/week), each for two weeks sequentially. For the remaining 46 weeks, patients will continue to receive MOD-4023 at a dose of 0.66 mg/kg/week.
  Interventions: Drug: MOD-4023
- Genotropin Treatment Arm (Active Comparator): Genotropin® (reference treatment): daily Genotropin® (0.025 mg/kg/day).
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: MOD-4023 — MOD-4023 is a long-acting modified recombinant human growth hormone (r-hGH) which utilizes C-terminal peptide (CTP) technology. It will be provided as a solution for injection containing 20 or 50 mg/mL MOD-4023 in a multi-dose disposable pre-filled PEN.
  MOD-4023 will be administered as a SC injection once weekly, using a delivery device.
  Other Names: Somatrogon
  Arms: MOD-4023 Treatment Arm
Drug: Genotropin — Genotropin® is dispensed in a 2-chamber cartridge. The front compartment contains recombinant somatropin, glycine, mannitol, sodium dihydrogen phosphate anhydrous and disodium phosphate anhydrous. The rear compartment contains m-Cresol and mannitol in water for injections.
  A delivery device (Genotropin®) will be used for daily (evening/bedtime) SC administration of Genotropin® into the region of the upper arms, buttocks, thighs or abdomen (8 locations). Injection sites should be rotated.
  Dose regimen for Genotropin®: 0.025 mg/kg/day (or 0.175 mg/kg/w divided equally to 7 injections over a week).
  Arms: Genotropin Treatment Arm

SUMMARY:
Treatment of children with growth failure due to growth hormone deficiency (GHD).

Primary • To evaluate the efficacy and safety of weekly MOD-4023 administration compared to daily Genotropin® administration in Japanese pre-pubertal children with GHD.

Secondary

• To evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) profiles of three different doses of MOD-4023 in Japanese pre-pubertal children with GHD.

DETAILED DESCRIPTION:
This is a 12-month, open-label, randomized, active controlled, parallel group study comparing the efficacy and safety of weekly MOD-4023 to daily recombinant human growth hormone (r-hGH), Genotropin ®. Both drugs will be injected subcutaneously (SC) using a pen device.

After a 4 week Screening period, patients meeting all the entry criteria and none of the exclusion criteria, will be eligible to participate in the study.

Eligible patients will be randomized in a 1:1 ratio, to receive either:

• MOD-4023 (investigational treatment): weekly MOD-4023 SC injections for 12 months; initially over the first 6 weeks, MOD-4023 will be administered in 3 stepwise escalating doses (0.25 mg/kg/week, 0.48 mg/kg/week and 0.66 mg/kg/week), each for two weeks sequentially. For the remaining 46 weeks, patients will continue to receive MOD-4023 at a dose of 0.66 mg/kg/week.

Or

• Genotropin® (reference treatment): daily Genotropin® (0.025 mg/kg/day which is equivalent to 0.175 mg/kg/week, divided equally into 7 daily injections over a week) SC injection for 12 months.

After the 6-week PK/PD sampling period, the dose of MOD-4023 and Genotropin® will be adjusted every 3 months based on a patient's body weight. Doses may be decreased for safety reasons according to the pre-defined dose-adjustment criteria (which will be based on the severity of adverse events (AEs) or repeated, elevated levels of IGF-1 Standard Deviation Score (SDS)).

The key safety data will be reviewed by an independent and external Data and Safety Monitoring Board (DSMB). DSMB review will also include a review of the number or percentage of patients requiring dose reductions due to AEs. Following the completion of the12-month treatment period, eligible patients will be consented to enroll into an open-label long term extension (LTE) period, and an amendment to this study protocol will be submitted prior to the first patient completes the 12 months treatment period. Eligible Genotropin®-treated patients will be switched to a MOD-4023 dose of 0.66 mg/kg/week in the LTE. The LTE is planned to continue until MOD-4023 marketing registration in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-pubertal child aged ≥ 3 years old, and not yet 10 years for girls (9 years and 364 days) or not yet 11 years for boys (10 years and 364 days), on the date of ICF signature, with either isolated GHD, or GH insufficiency as part of multiple pituitary hormone deficiency.
2. Confirmed diagnosis of GHD by 2 different types of GH provocation tests (standardized on growth foundation data): defined as a peak serum GH level of ≤ 6.0 ng/mL or ≤ 16 ng/mL when conducting GHRP-2 provocation test.

   Prior local laboratory results will be accepted subject to pre-approval by the study medical monitor and if the tests were conducted as specified in the protocol.
3. Bone age (BA) is not older than chronological age and should be less than 10 for girls and less than 11 for boys.
4. Without prior exposure to any r-hGH therapy.
5. Height SD score ≤ -2.0 at screening
6. Impaired height velocity defined as:

   * Annualized height velocity (HV) below the 25th percentile for CA (HV < -0.7 SDS) and gender according to the local primary care provider standard.
   * The interval between two height measurements should be at least 6 months, but should not exceed 18 months prior to inclusion.
7. BMI must be within ±2 SDS of mean BMI for the chronological age and sex.
8. Baseline IGF-1 level of at least 1 SDS below the mean IGF-1 level standardized for age and sex (IGF-1 SDS ≤ -1) according to the central laboratory reference values. A single re-test will be allowed (subject to discussion with the study medical monitor) if all other criteria are met.
9. Normal creatinine levels according to common practice reference ranges per age.
10. Children with multiple hormonal deficiencies must be on stable replacement therapies (no change in dose) for other hypothalamo-pituitary organ axes for at least 3 months prior to ICF signing
11. Normal 46 XX karyotype for girls.
12. Willing and able to provide written informed consent of the parent or legal guardian of the patient and written assent from pediatric patients (when applicable based on age and Japan regulation).

Exclusion Criteria:

1. Children with prior history of leukemia, lymphoma, sarcoma or any other forms of cancer.
2. History of radiation therapy or chemotherapy
3. Malnourished children defined as BMI < -2 SDS for age and sex
4. Children with suspected psychosocial dwarfism by the discretion of the investigator
5. Children born small for gestational age (SGA - birth weight and/or birth length < -2 SDS for gestational age)
6. Presence of anti-hGH antibodies at screening
7. Any clinically significant abnormality likely to affect growth or the ability to evaluate growth, such as, but not limited to, chronic diseases like renal insufficiency, spinal cord irradiation, etc.
8. Children with diabetes mellitus
9. Chromosomal abnormalities including Turner's syndrome, Laron syndrome, Noonan syndrome, Prader-Willi syndrome, Russell-Silver syndrome, SHOX (short stature homeobox) mutations/deletions and skeletal dysplasia's, with the exception of septo-optic dysplasia.
10. Concomitant administration of other treatments that may have an effect on growth such as anabolic steroids, sex steroids, with the exception of ADHD drugs or hormone replacement therapies (thyroxin, hydrocortisone, desmopressin [DDAVP])
11. Children requiring glucocorticoid therapy (e.g. for asthma) that are taking chronically a dose greater than 400 µg/d of inhaled budesonide or equivalent as provided in Appendix J.
12. Major medical conditions and/or presence of contraindication to r-hGH treatment.
13. Known or suspected HIV-positive patient, or patient with advanced diseases such as AIDS or tuberculosis.
14. Drug substance or alcohol abuse.
15. Known hypersensitivity to the components of study medication.
16. Other causes of short stature such as celiac disease, uncontrolled primary hypothyroidism and rickets.
17. The patient and/or the parent/legal guardian are likely to be non-compliant in respect to study conduct.
18. Participation in any other clinical trial within 30 days prior to screening and throughout the entire study period (including administration of investigational agent).

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Pre-pubertal child aged ≥ 3 years old, and not yet 10 years for girls (9 years and 364 days) or not yet 11 years for boys (10 years and 364 days), on the date of ICF signature.
Enrollment: 44 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reiko Horikawa, M.D, Ph. D., Principal Investigator — National Center for Child Health and Development
Locations (46):
- Japan (46):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Seirei Sakura Citizen Hospital, Sakura, Chiba
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - National Hospital Organization Kure Medical Center & Chugoku Cancer Center, Kure, Hiroshima
  - Onomichi General Hospital, Onomichi, Hiroshima
  - Hokkaido P.W.F.A.C. Asahikawa-Kosei General Hospital, Asahikawa, Hokkaido
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - KKR Sapporo Medical Center, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Takahashi Clinic, Kobe, Hyōgo
  - Takarazuka City Hospital, Takarazuka, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto
  - East Japan Railway Company Sendai Branch Office JR Sendai Hospital, Sendai, Miyagi
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai, Miyagi
  - Igarashi childrens clinic, Sendai, Miyagi
  - Oita University Hospital, Yufu, Oita Prefecture
  - Osaka Women's and Children's Hospital, Izumi, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical University Hospital, Iruma-Gun, Saitama
  - Saitama Medical Center, Kawagoe, Saitama
  - Shimane University Hospital, Izumo, Shimane
  - Tokyo Metropolitan Childrens Medical Center, Fuchū, Tokyo
  - National Center for Child Health and Development, Setagaya-Ku, Tokyo
  - Keio University Hospital, Shinjuku, Tokyo
  - Teikyo University Hospital, tabashi City, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Akita University Hospital, Akita
  - Fukuoka Children's Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima City Hospital Organization Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Kumamoto University Hospital, Kumamoto
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki
  - Arakawa Children's Clinic, Nagano
  - Nara Prefecture General Medical Center, Nara
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama Saiseikai General Hospital Outpatient Center, Okayama
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Saitama Childrens Medical Center, Saitama
  - Saitama City Hospital, Saitama
  - Shizuoka Childrens Hospital, Shizuoka
  - Toranomon Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horikawa R, Tanaka T, Hasegawa Y, Yorifuji T, Ng D, Rosenfeld RG, Hoshino Y, Okayama A, Ebata N, Hosoi M, Nakamuta S, Gomez R, Pastrak A, Castellanos O. Efficacy and safety of once-weekly somatrogon following up to 4 years of treatment in Japanese children with growth hormone deficiency: results from an open-label extension of a phase 3 study. Endocr J. 2025 Oct 31. doi: 10.1507/endocrj.EJ24-0625. Online ahead of print. PMID 41183961

RESULTS

PARTICIPANT FLOW:
Groups:
- MOD-4023 Treatment Arm: MOD-4023 (investigational treatment): weekly MOD-4023 SC injections for 12 months; initially over the first 6 weeks, MOD-4023 will be administered in 3 stepwise escalating doses (0.25 mg/kg/week, 0.48 mg/kg/week and 0.66 mg/kg/week), each for two weeks sequentially. For the remaining 46 weeks, patients will continue to receive MOD-4023 at a dose of 0.66 mg/kg/week.
  MOD-4023: MOD-4023 is a long-acting modified recombinant human growth hormone (r-hGH) which utilizes C-terminal peptide (CTP) technology. It will be provided as a solution for injection containing 20 or 50 mg/mL MOD-4023 in a multi-dose disposable pre-filled PEN.
  MOD-4023 will be administered as a SC injection once weekly, using a delivery device.
- Genotropin Treatment Arm: Genotropin® (reference treatment): daily Genotropin® (0.025 mg/kg/day).
  Genotropin: Genotropin® is dispensed in a 2-chamber cartridge. The front compartment contains recombinant somatropin, glycine, mannitol, sodium dihydrogen phosphate anhydrous and disodium phosphate anhydrous. The rear compartment contains m-Cresol and mannitol in water for injections.
  A delivery device (Genotropin®) will be used for daily (evening/bedtime) SC administration of Genotropin® into the region of the upper arms, buttocks, thighs or abdomen (8 locations). Injection sites should be rotated.
  Dose regimen for Genotropin®: 0.025 mg/kg/day (or 0.175 mg/kg/w divided equally to 7 injections over a week).
Period: Overall Study
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: Year] | 5.28 (1.84) | 6.78 (2.34) | 6.03 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 9 | 12 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  Japan | 22 | 22 | 44
Weight (kilogram) [Mean (Standard Deviation); unit: Kilogram] | 14.49 (3.33) | 17.87 (4.85) | 16.18 (4.45)
Body mass index (kilogram/meter^2) [Mean (Standard Deviation); unit: Kilogram/meter^2] | 15.27 (1.30) | 15.89 (1.09) | 15.58 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: Annual Height Velocity (HV) After 12 Months
Description: Annual Height Velocity in cm/year after 12 months of treatment.
Time Frame: 12 months
Population: One subject in the Genotropin arm did not finish the 12 month period and therefore not included in primary outcome.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm
Number analyzed (Participants) | 22 | 21
cm/year | 9.78 (1.59) | 7.78 (1.14)

2. Secondary Outcome: Height Velocity at 6 Months
Description: Annualized height velocity (cm/year) for the MOD-4023 and the daily hGH treatment groups
Time Frame: 6 months
Population: One subject in the Genotropin arm was discontinued from treatment before the 6 month period and therefore not included in secondary outcome.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm
Number analyzed (Participants) | 22 | 21
cm/year | 10.54 (2.04) | 8.34 (1.84)

3. Secondary Outcome: Change in Height Standard Deviation Score (SDS) Compared to Baseline After 12 Months
Description: Change in height standard deviation score (SDS) for the MOD-4023 and the daily hGH treatment groups
  Height Standard Deviation Score (SDS) is the number of standard deviations above or below the mean height for age and sex. Height in cm is converted to height standard deviation score (SDS) by subtracting the mean and dividing by the SD. A higher Height Standard Deviation Score (SDS) indicates a better outcome
Time Frame: 12 months
Population: One subject in the Genotropin arm did not finish the 12 month period and therefore not included in secondary outcome.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm
Number analyzed (Participants) | 22 | 21
Standard Deviation Score (SDS) | 0.97 (0.41) | 0.50 (0.23)

4. Secondary Outcome: Change in Bone Maturation (BM) After 12 Months
Description: Change in bone maturation (bone age / chronological age) with the method of TW2 using a central bone age reader.
Time Frame: 12 months
Population: One subject in the Genotropin arm did not finish the 12 month period and therefore not included in secondary outcome.
Measure: Mean (Standard Deviation); unit: ratio of bone age to chronologic age
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm
Number analyzed (Participants) | 22 | 21
ratio of bone age to chronologic age | 0.05 (0.06) | 0.03 (0.06)

5. Other Pre Specified Outcome: Biochemical
Description: IGF-1 Standard Deviation Score on day 4(-1) after MOD-4023 dosing across study visits (window only applies to visits 6 to 9)
  Height Standard Deviation Score (SDS) is the number of standard deviations above or below the mean height for age and sex. Height in cm is converted to height standard deviation score (SDS) by subtracting the mean and dividing by the SD. A higher Height Standard Deviation Score (SDS) indicates a better outcome
Time Frame: Baseline, Visit 6 (Month 3), Visit 7 (Month 6), Visit 8 (Month 9) and Visit 9 (12 months)
Population: One subject in the Genotropin group dropped out due to AE, so no data for 6 and 9 months.
Measure: Median (Standard Deviation); unit: Standard Deviation Score
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm
Number analyzed (Participants) | 22 | 22
Standard Deviation Score
  Baseline | -1.460 (0.902) | -1.420 (0.843)
  Visit 6 (Month 3) | 0.960 (0.770) | -0.620 (0.744)
  Visit 7 (Month 6): number analyzed (Participants) | 22 | 21
  Visit 7 (Month 6) | 1.055 (0.834) | -0.130 (0.725)
  Visit 8 (Month 9): number analyzed (Participants) | 22 | 21
  Visit 8 (Month 9) | 1.465 (0.953) | -0.310 (0.951)
  Visit 9 (Month 12) | 1.435 (0.921) | -0.855 (1.077)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Genotropin Treatment Arm: Genotropin® (reference treatment): daily Genotropin® (0.025 mg/kg/day).
  Genotropin: Genotropin® is dispensed in a 2-chamber cartridge. The front compartment contains recombinant somatropin, glycine, mannitol, sodium dihydrogen phosphate anhydrous and disodium phosphate anhydrous. The rear compartment contains m-Cresol and mannitol in water for injections.
  A delivery device (GenotropinÒ) will be used for daily (evening/bedtime) SC administration of Genotropin® into the region of the upper arms, buttocks, thighs or abdomen (8 locations). Injection sites should be rotated.
  Dose regimen for Genotropin®: 0.025 mg/kg/day (or 0.175 mg/kg/w divided equally to 7 injections over a week).
Arm/Group | MOD-4023 Treatment Arm | Genotropin Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/22 | 2/22
Other Adverse Events (participants affected / at risk) | 22/22 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 Treatment Arm (N=22) | Genotropin Treatment Arm (N=22)
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Febrile convulsion (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 Treatment Arm (N=22) | Genotropin Treatment Arm (N=22)
Conjunctivitis allergic (Eye disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Injection site erythema (General disorders) | 2 | 0
Injection site pain (General disorders) | 16 | 3
Pyrexia (General disorders) | 4 | 3
Bronchitis (Infections and infestations) | 4 | 1
Conjunctivitis (Infections and infestations) | 1 | 5
Erythema infectiosum (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 4 | 2
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 6 | 6
Nasopharyngitis (Infections and infestations) | 12 | 11
Otitis media (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 3 | 4
Rhinitis (Infections and infestations) | 2 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT03874013/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03874013/SAP_001.pdf